CLINICAL TRIAL: NCT05059470
Title: IMRT Followed by Pembrolizumab in the Adjuvant Setting in Anaplastic Cancer of the Thyroid (IMPAACT): Phase II Trial Adjuvant Pembrolizumab After IMRT in ATC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: <75% participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0704; NCI-2021-10669 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2021-09-15; First posted 2021-09-28 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab (Experimental): The infusions are given every 6 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Given by IV

SUMMARY:
This is an open label, single center, phase 2 trial of adjuvant pembrolizumab after external beam radiation to the primary tumor in patients with stage IVB (disease localized to the neck) ATC. This drug trial will estimate the median progression-free survival (PFS) (from the start of adjuvant pembrolizumab until locoregional progression, development of distant metastatic disease, or death) in stage IVB ATC patients with gross disease, treated with external beam radiation (+/- concomitant chemotherapy) followed by adjuvant pembrolizumab. Patients will be patients enrolled from cohort 1 and 2 (cohort 1: ≥51 Gy; cohort 2: ≤50 Gy).

DETAILED DESCRIPTION:
Primary Objective:

-To estimate the median progression-free survival (PFS) (from the start of adjuvant pembrolizumab until locoregional progression, development of distant metastatic disease, or death) in stage IVB ATC patients with gross disease, treated with external beam radiation (+/- concomitant chemotherapy) followed by adjuvant pembrolizumab. Patients will be patients enrolled from cohort 1 and 2 (cohort 1: ≥51 Gy; cohort 2: ≤50 Gy).

Secondary Objective:

-To estimate median overall survival in stage IVB ATC patients treated with external beam radiation (+/- concurrent chemotherapy) followed by adjuvant pembrolizumab. Patients will be stratified by dose of external beam radiation.

Exploratory Objective:

-To estimate the median disease-free survival (DFS) in patients with stage IVB ATC treated with surgery/external beam radiation/concomitant chemotherapy followed by adjuvant pembrolizumab (cohort 3).

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with Pathologic findings supporting the clinical impression of anaplastic thyroid carcinoma will be enrolled in this study. Diagnosis may include consistent with or suggestive of terminology associated with: anaplastic thyroid carcinoma, undifferentiated carcinoma, squamous carcinoma; carcinoma with spindled, giant cell, or epithelial features; poorly differentiated carcinoma with pleomorphism, extensive necrosis with tumor cells present.
2. Stage IVB disease (no convincing evidence of metastatic disease outside of the neck) who have unresectable disease are eligible in groups 1 or 2. Previous excisional biopsy is permitted.
3. Stage IVB disease (no convincing evidence of metastatic disease outside of the neck) who have undergone complete resection of tumor (no convincing evidence of metastatic disease in the neck) are eligible in group 3
4. Patient must have completed external beam radiation with or without concomitant cytotoxic chemotherapy to participate in groups 1 and 2. Those who have completed these treatment after surgical resection of primary tumor may participate in group 3.
5. Patients may enroll only after completing radiation. Study drug may start from 2-6 weeks (+2 weeks) after radiation is completed and can only be started once radiation and chemotherapy-related toxicities are grade 2 or less (with the exception of alopecia). If a subject is consented but AEs are not grade 2 or less by 8 weeks after RT is completed, that subject is not eligible and should not start pembrolizumab.
6. A female participant is eligible to participate if she is not pregnant (see Appendix 3), not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP) as defined in Appendix 3 OR
   2. A WOCBP who agrees to follow the contraceptive guidance in Appendix 3 during the treatment period and for at least 120 days after the last dose of study treatment.
7. A male participant must agree to use a contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 32 weeks (5 terminal half-lives for pembrolizumab plus an additional 90 days) from the last dose of study treatment and refrain from donating sperm during this period.
8. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days prior to the first dose of study intervention.
10. Adequate organ function as defined in the following table (Table 1). Specimens must be collected within 10 days prior to the start of study intervention.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to first dose of pembrolizumab (see Appendix 3). A serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
3. Has received a live vaccine or live-attenuated vaccine within 30 days prior to the first dose of study drug. Administration of killed vaccines is allowed.
4. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention.
5. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
6. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
7. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
8. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease, not related to radiation.
9. Has an active infection requiring systemic therapy.
10. Has a known history of Human Immunodeficiency Virus (HIV) infection.
11. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as HCV RNA qualitative is detected) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-02-11 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
To establish the median progression-free survival (PFS). | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cabanillas, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2023-04-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT05059470/ICF_000.pdf